CLINICAL TRIAL: NCT06623708
Title: SMARTCLOTH. Design, Implementation and Study of the Effectiveness and Usability of a Digital Tablecloth for Self-management of Diet in Diabetic Patients.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI21/01602
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus Type 2; Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This group of participants should follow the general recommendations for the management of Type 1 or Type 2 Diabetes.
- SMARTCLOTH (Experimental): This group will use SMARTCLOTH for 3 months.
  Interventions: Device: SMARTCLOTH

INTERVENTIONS:
Device: SMARTCLOTH — The intervention consists of using SMARTCLOTH. This device makes it possible to monitor dietary intake throughout the day and record it in a database that, through a website, allows to track it. SMARTCLOTH is a digital tablecloth consisting of a scale, several buttons and a screen. The device allows weighing the food to be consumed and recording its nutritional value (macronutrients in grams, macronutrient servings and kilocalories). The latter is achieved because SMARTCLOTH allows the patient to select to which food group the food being weighed belongs, increasing the accuracy of the nutritional estimation.
  Arms: SMARTCLOTH

SUMMARY:
The objective of this clinical trial is to know the usability and efficacy of SMARTCLOTH for better control and adherence to the dietary patterns recommended to patients with diabetes, both the portion diet system (more common for cases of Diabetes Mellitus type 1 -DM1-), and the plate method (more recommended in cases of Diabetes Mellitus type 2-DM2-). The main questions are:

* Does the use of SMARTCLOTH improve glycemic control in patients with diabetes mellitus?
* Do patients with diabetes mellitus find SMARTCLOTH useful in their daily lives?

The researchers will compare changes over 3 months in variables related to glycemic control in two groups, one using SMARTCLOTH (intervention group) and the other following standard recommendations (control group). To do so, participants will have to:

* Use SMARTCLOTH for 3 months or follow the recommendations they receive from their referring health professionals.
* Come back after three months for a check-up of the chosen variables.
* The experimental group should contact the investigators in case the hardware has any problems.

ELIGIBILITY:
Inclusion Criteria: Subjects with type 1 and 2 diabetes (eligible population) aged between 18 and 70 years with disease progression not exceeding 15 years and HbA1c greater than 7.5.

Exclusion Criteria:

* Degree of dependence (physical or psychological) that makes it impossible for them to perform autonomous self-care of the dietary-nutritional regimen.
* Oncological or autoimmune disease, chronic renal insufficiency, transplant patients and others that alter the values of the result variables or may constitute a confounding factor.
* Other diseases that entail surgical interventions or hospital admissions that make it impossible to follow up the study.
* Patients with complications due to the evolution of the diabetic pathology: retinopathy, nephropathy, polyneuropathy, ischemic heart disease, as well as other micro and macrovascular complications derived from the same and already recorded in the patient.
* Those subjects subjected to specific dietary regimes such as celiac disease, lactose intolerant, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
glycated hemoglobin | From enrollment to the end of treatment at 3 months
  The test shows an average of the blood sugar level over the past 90 days and represents a percentage. The test can also be used to diagnose diabetes

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Ugc Centro, Córdoba, Andalusia
  - Ugc Lucano, Córdoba, Andalusia
  - Ugc Aeropuerto, Córdoba, Andalusia
  - Ugc Fuensanta, Córdoba, Andalusia
  - Ugc La Carlota, Córdoba, Andalusia

IPD SHARING:
Plan to Share IPD: No